CLINICAL TRIAL: NCT05143190
Title: A Phase 2b Open-Label Study of PTR-01 in Recessive Dystrophic Epidermolysis Bullosa (RDEB) Patients Previously Treated With PTR-01 in Study PTR-01-002
Brief Title: Extension Study to PTR-01-002 (A Study in Recessive Dystrophic Epidermolysis Bullosa (RDEB) Patients Previously Treated With PTR-01)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phoenix Tissue Repair, Inc. (Industry)
Collaborators: Phoenix Tissue Repair, a BridgeBio company (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTR-01-003
Record Dates: First submitted 2021-11-09; First posted 2021-12-03 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Recessive Dystrophic Epidermolysis Bullosa
Keywords: Dystrophic Epidermolysis Bullosa; Epidermolysis Bullosa; RDEB; EB
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa

STUDY DESIGN:
Intervention Model Description: Phase 2 open-label
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PTR-01 (Experimental): All patients will receive a PTR-01 dose of 3.0 mg/kg once weekly every week for a total of 4 doses, followed by a dose of 3.0 mg/kg once monthly for a total of 5 doses.
  Interventions: Drug: PTR-01

INTERVENTIONS:
Drug: PTR-01 — Intravenous recombinant collagen 7
  Other Names: Recombinant collagen 7 (rC7)

SUMMARY:
A sub-set of patients who participated in PTR-01-002 will be enrolled in an open-label study, if they meet the study eligibility criteria.

DETAILED DESCRIPTION:
Protocol PTR-01-003 is a 4-part Phase 2, open-label study of PTR-01 in patients who satisfactorily completed study PTR-01-002 and meet current enrollment criteria.

In Part 1, patients will be monitored monthly for up to 2 months with patient-reported and Investigator assessments. In Part 2, patients will receive a dose of 3.0 mg/kg every week for a total of 4 doses. This will be followed by Part 3 in which patients will receive a dose of 3.0 mg/kg monthly for a total of 5 additional doses. At the end of each dosing period, efficacy assessments will be performed. During Part 4, patients will be evaluated at Months 1 and 3 after completion of dosing to assess the durability of wound healing and other efficacy parameters. Safety will be assessed continuously throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide informed consent form, or if 12 to <18 years of age, legal guardian has provided informed consent form and the minor has signed an assent form acknowledging that they understand and agree to study procedures.
2. Has satisfactorily completed participation in PTR-01-002.
3. Agrees to use contraception as follows:

   * For women of childbearing potential (WOCBP) agrees to use highly effective contraceptive (including abstinence) methods from Screening, through the study, and for at least 10 weeks after the last dose of study drug. Non-childbearing potential is defined as a female who meets either of the following criteria: age ≥50 years and no menses for at least 1 year or documented hysterectomy, bilateral tubal ligation, or bilateral oophorectomy.
   * For males, agrees to use a condom with any WOCBP sexual partner from Day 1 of study treatment, through the study, and at least 10 weeks after the last dose of study drug.
4. Be willing and able to comply with this protocol.

Exclusion Criteria:

1. Has known systemic hypersensitivity to any of the inactive ingredients in PTR-01.
2. Has previously had an anaphylactic reaction to PTR-01.
3. Is pregnant or nursing.
4. Has received in the last six months any investigational gene therapy product or in the last three months any non-gene therapy investigational products (other than PTR-01).
5. Is anticipated to receive new regimens of antibiotics or other anti-infectives during the trial.
6. Has any other medical or personal condition that, in the opinion of the Investigator, may potentially compromise the safety or compliance of the

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Sustained wound healing | Up to 246 days
  Change in a majority of target lesions of at least 2 levels using a 7-point (1-7) Global Impression of Change instrument (7 being the worst)
Incidence of treatment-emergent adverse events | Up to 246 days
  Safety and tolerability, as assessed by treatment-emergent adverse events

SECONDARY OUTCOMES:
Delivery of recombinant collagen 7 (PTR-01) to skin | Up to 246 days
  Amount of recombinant collagen 7 (PTR-01) incorporation to skin as compared to normal human skin assessed by immunofluorescence using NC1 & NC2 antibody staining
Formation of anchoring fibrils | Up to 246 days
  Formation of new anchoring fibrils as measured by electron microscopy
Change in wound surface area | Up to 246 days
  Wound surface area of lesions as assessed by medical photography using the Canfield RUBI 3D imaging system
Change in skin integrity, as assessed by suction blister time | Up to 246 days
  Change in skin integrity, as assessed by suction blister time
Change in skin integrity, as assessed by time to re-blistering | Up to 246 days
  Change in skin integrity, as assessed by time to re-blistering
Change in itch severity, as assessed by modified Patient-Reported Outcome Measurement Information System (PROMIS) itch domains | Up to 246 days
  Severity of itch, as assessed by modified Patient-Reported Outcome Measurement Information System (PROMIS) itch domains, maximum score of 5 (worst)
Change in the impact of itch on quality of life | Up to 246 days
  Change in the impact of itch on quality of life, as assessed by the Pruritus-Specific Quality of Life Instrument (ItchyQoL), maximum score of 110 (worst)
Change in pain severity, as assessed by modified Patient-Reported Outcome Measurement Information System (PROMIS) pain domains | Up to 246 days
  Change in pain severity, as assessed by Patient-Reported Outcome Measurement Information System (PROMIS) pain domains, maximum score of 5 (worst)
Change in pain severity, as assessed by the Instrument for Scoring Clinical Outcomes for Research of Epidermolysis Bullosa (iscorEB) | Up to 246 days
  Change in pain severity, as assessed by the Instrument for Scoring Clinical, maximum score of 234 (worst)
Change of dysphagia, as assessed using the Brief Esophageal Dysphagia Questionnaire | Up to 246 days
  Change of dysphagia, as assessed using the Brief Esophageal Dysphagia Questionnaire, maximum score is 40 (worst)
Stabilization of dysphagia, as assessed using the Brief Esophageal Dysphagia Instrument | Up to 246 days
  Stabilization of dysphagia, as assessed using the Brief Esophageal Dysphagia Instrument, maximum score of 40 (worst)
Change in corneal symptoms | Up to 246 days
  Change of corneal symptoms (eye symptoms), as assessed by the Epidermolysis Bullosa Eye Disease Index (EB-EDI), maximum score of 100 (worst)
Stabilization of corneal symptoms | Up to 246 days
  Stabilization of corneal symptoms (eye symptoms), as assessed by the Epidermolysis Bullosa Eye Disease Index (EB-EDI), maximum score of 100 (worst)
Rate of change in nutritional markers (hemoglobin) | Up to 246 days
  Change of nutritional markers, as assessed by hemoglobin
Rate of change in nutritional markers (hematocrit) | Up to 246 days
  Change of nutritional markers, as assessed by hematocrit
Rate of change in nutritional markers (total protein/albumin) | Up to 246 days
  Change of nutritional markers, as assessed by total protein/albumin
Rate of change in nutritional markers (Fe/TIBC) | Up to 246 days
  Change of nutritional markers, as assessed by total Fe/TIBC
Rate of change in nutritional markers (C-reactive protein) | Up to 246 days
  Change of nutritional markers, as assessed by total C-reactive protein
Change in Investigator Global Impressions of Change (IGIC) | Up to 246 days
  Global impressions of change, as assessed through IGIC (1-7), 7 being worst
Change in Investigator Patient Impressions of Change (PGIC) | Up to 246 days
  Global impressions of change, as assessed through PGIC (1-7), 7 being worst
Change in overall quality of life, as assessed by the Quality of Life in Epidermolysis Bullosa (QOLEB) questionnaire | Up to 246 days
  Change in overall quality of life, as assessed by the Quality of Life in Epidermolysis Bullosa (QOLEB) questionnaire maximum score is 67 (worst)
Change in overall health | Up to 246 days
  Change in overall disability, as assessed by the Health Assessment Questionnaire or Children's Health Assessment Questionnaire (HAQ/CHAQ) maximum score is 3 (worst)
Change in mental health | Up to 246 days
  Change in mental health, as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) mental health domains, maximum score is 5 (worst)
Change in social function | Up to 246 days
  Change in social functioning, as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) social function domains, maximum score is 4 (worst)
Change in amount of wound care | Up to 246 days
  Change in amount of wound care, as assessed by patient interviews
Change in time for wound care | Up to 246 days
  Change in time for wound care, as assessed by patient interviews
Change in cost of wound care | Up to 246 days
  Change in cost of wound care, as assessed by patient interviews
Change in overall patient impression of quality of life | Up to 246 days
  Change in overall anecdotal quality of life, as assessed by one-on-one patient interviews
Change in overall patient impression of disability | Up to 246 days
  Change in overall anecdotal disability, as assessed by one-on-one patient interviews
Effect of anti-drug antibodies (ADA) on pharmacokinetics parameter Cmax | Up to 246 days
  Correlate ADA with Cmax
Effect of anti-drug antibodies (ADA) on pharmacokinetics parameter Tmax | Up to 246 days
  Correlate ADA with Tmax
Effect of anti-drug antibodies (ADA) on pharmacokinetics parameter Area Under the Curve (AUC) | Up to 246 days
  Correlate ADA with Area Under the Curve (AUC)
Effect of anti-drug antibodies (ADA) on pharmacokinetics parameter of clearance of PTR-01 | Up to 246 days
  Correlate ADA with clearance of PTR-01
Effect of anti-drug antibodies (ADA) on pharmacokinetics parameter of PTR-01 half-life | Up to 246 days
  Correlate ADA with PTR-01 half-life

CONTACTS AND LOCATIONS:
Overall Officials: Dan Rudin, MD, Study Director — Phoenix Tissue Repair
Locations (2):
- United States (2):
  - Stanford University, Redwood City, California
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No